CLINICAL TRIAL: NCT03810781
Title: Study of Postural Stability in Subjects With Myelopathy Using a Portable Virtual Reality Balance Protocol
Brief Title: Postural Stability in Cervical Spinal Myelopathy
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: F2882-P; RX002882-01A1 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Cervical Spondylotic Myelopathy
Keywords: Posturography; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cervical Spondylotic Myelopathy (CSM): Degenerative cervical myelopathy, encapsulates a cascade of events leading to significant degenerative changes in discs, formation of osteophytes, facet hypertrophy, calcification of the posterior longitudinal ligament and ligamentous flavum with resultant canal stenosis and segmental instability.

SUMMARY:
Veterans are at heightened risk of developing cervical spondylotic myelopathy (CSM) from rigors of military service. Balance and posturography are negatively affected in CSM, but require expensive equipment, and extensive training of personnel for data acquisition and interpretation. The Virtual Environment TBI Screen (VETS) is a simple and inexpensive construct that could be implemented as an aid in diagnosis and as an objective means to compare treatment modalities and track recovery. The goal for the SPiRE is to generate the critical data to support rigorous Merit studies of posturography for assessments of clinical course in the treatment and rehabilitation of CSM. The investigators' ultimate goal, if the SPiRE is successful, is to phase in objective posturography assessments as VA standard of care in CSM.

DETAILED DESCRIPTION:
COVID-19 administrative hold

Veterans are at heightened risk of developing cervical spondylotic myelopathy (CSM) from rigors of military service. Diagnosis of CSM involves a set of clinical findings and is confirmed by imaging the spine.

Gait impairment and disturbances of stance control are hallmarks of CSM and are a consequence of abnormalities in proprioception due to dorsal column tract damage of the spine. Currently, gait and balance deficits rely on clinical level assessments and judgement for detection. An objective measure of posturography has the benefit of: a) quantifying balance-related disability in CSM, b) facilitating structure-functional assessments in CSM, and c) quantifying the degree surgical interventions affect posturography and recovery of function in CSM.

Objective and sensitive means for assessing balance and posturography exist, but are not routinely incorporated in diagnosis or functional tracking of progress after interventions such as surgery. A barrier may be accessibility of posturography and ease of assessments. The Virtual Environment TBI Screen (VETS) was devised using Army Rapid Innovation Development funding to objectively assess balance and posturography in a cost effective, but sensitive manner. VETS involves virtual environments and computerized posturography and is proving to be a sensitive system facilitating diagnosis, treatment, and mitigation of balance dysfunction associated with mTBI.

The working hypothesis is VETS testing will enhance clinical judgements regarding CSM. The SPiRE is designed to provide data critical to a more extensive program of research incorporating posturography into treatment and rehabilitation of CSM.

First, a limited comparative study of standing balance will be conducted of 20 Veterans being evaluated for cervical spine surgery to treat CSM and 20 otherwise healthy Veterans. Second, posturography of the Veterans undergoing surgery to treat CSM will be tracked during their scheduled follow up visits to determine the degree VETS scores are affected by surgery and to track recovery from CSM.

Patients in the CSM group will be selected based on clinical criteria. Veterans in the control group will be recruited from the Syracuse Veterans Affairs Medical Center (SVAMC) and surrounding community.

For VETS testing, the Veteran will stand directly on a firm surface or foam pad placed on top of a Wii Balance Board (WBB). There are six conditions manipulating surface (firm or foam surface) and visual input (eyes open viewing a static scene, eyes closed, and eyes open viewing a dynamic visual scene). The primary measure is the center of pressure (COP) sway area. These 6 conditions allow for an assessment of generalized vs specific deficits in COP sway area considering proprioception, dependence of visual input and visuo-proprioceptive integration.

AIM 1A: Determine whether and to what degree balance is altered in CSM. The degree of COP sway will be compared between CSM and controls in the six conditions comprising VETS testing.

AIM 1B: Determine whether VETS enhances sensitivity and selectivity in the diagnosis of CSM. Composite measures of balance will be related to clinical assessment tools and their relationship with MRI.

AIM 2: Evaluate the VETS scores after surgery to treat CSM. The degree of COP sway area under the 6 conditions will be compared before surgery, 2 weeks, 6 weeks and 6 months after surgery (corresponding with post-operative clinical assessments).

The ultimate goal is to validate and incorporate objective balance testing into routine assessment for CSM to aid in disambiguating CSM, to improve functional assessments of recovery, and to aid in evaluations of different treatment and rehabilitation strategies in CSM for the Veteran population.

ELIGIBILITY:
Inclusion Criteria:

Patients in the CSM group will be selected based on clinical criteria. Inclusion criteria for the CSM group are:

* symptoms of myelopathy in upper and lower extremities and stenosis of the cervical spine demonstrated by MRI or myelography
* lower extremity muscle strength of 4 as quantified by manual muscle test (MMT) 36 or above
* ability to stand without support with eyes closed for 30 s or more
* Veterans in the control group will be recruited from the SVAMC and surrounding community using printed advertisements

Exclusion Criteria:

Exclusion criteria for all study participants are:

* presence of lower extremity or lumbar spine disease
* peripheral neuropathy
* history of other neurological disorder
* inability to stand in an upright position with both feet together and eyes closed
* Although the SVAMC population is predominately Caucasian and male, every effort will be made to recruit minorities and women
* The proposed study will neither target for recruitment nor will the investigators exclude pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US Veterans.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Servatius, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was significantly hampered by COVID-19 and research shut-downs. Myelopathy surgeries were significantly limited because of COVID as well. Participants were recruited from the pool of eligible individuals undergoing surgery for myelopathy in the Syracuse VA. Recruitment occurred between 2/7/19 and 7/26/22
Pre-assignment Details: This did not occur
Period: Overall Study
Arm/Group | Cervical Spondylotic Myelopathy (CSM)
Started | 8
Completed | 6 (Facility entrance constraints due to COVID shut down research completely, which led to some enrolled patients not continuing with the study. Three CSM participants did not complete some interventions during the six weeks and six months Post-op follow-up session.)
Not Completed | 2
Not completed — COVID shut down | 2

BASELINE CHARACTERISTICS:
Groups:
- Cervical Spondylotic Myelopathy (CSM) Group: Veterans with CSM. CSM is degenerative cervical myelopathy, encapsulates a cascade of events leading to significant degenerative changes in discs, formation of osteophytes, facet hypertrophy, calcification of the posterior longitudinal ligament and ligamentous flavum with resultant canal stenosis and segmental instability.
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (3.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Virtual Environment TBI System (VETS) Assessment of Static Posturography
Description: The postural stability task involves six conditions during which Veterans are instructed to look straight ahead and maintain an upright stance as stably as possible. Veterans are barefooted with feet comfortably placed ~25 cm apart. The six conditions are (1) Eyes Open (EO) Firm (2) Eyes Closed (EC) Firm, (3) Dynamic Scene (DYN) Firm, (4) EO Foam, (5) EC Foam, and (6) DYN Foam. a) Comparison of CSM vs. Control and within-subject visual (EO,EC, and DYN) and surface conditions (FIRM and FOAM). b) Comparison of balance and posture at Pre-surgery for CSM group to age and gender matched non-CSM controls. Only pre-surgery data in CSM group was collected due to COVID-19.
Time Frame: Pre-Surgery compared to otherwise healthy Veterans
Population: COVID facility entry restrictions at the Syracuse VA Medical Center prevented the recruitment of participants who were not already coming to the VA for medical appointments.
Measure: Mean (Standard Deviation); unit: Square Centimeters
Groups:
- Pre-surgical Group: Cervical Spondylotic Myelopathy (CSM): Pre-surgical group: Degenerative cervical myelopathy, encapsulates a cascade of events leading to significant degenerative changes in discs, formation of osteophytes, facet hypertrophy, calcification of the posterior longitudinal ligament and ligamentous flavum with resultant canal stenosis and segmental instability.
- Healthy Controls: Control participants with no spinal problems
Arm/Group | Pre-surgical Group: Cervical Spondylotic Myelopathy (CSM) | Healthy Controls
Number analyzed (Participants) | 6 | 0
Square Centimeters
  EO Firm | 11 (27.1) |
  EC Firm | 13.0 (15.4) |
  DYN Firm | 48.4 (51.1) |
  EO Foam | 19.1 (20.3) |
  EC Foam | 44 (32.7) |
  DYN Foam | 70.7 (47.7) |

2. Primary Outcome: Change in Static Posturography (VETS)
Description: The Pre-surgery CSM group recruited for VETS (Static Posturography) measurement will also serve as the sample for the change in VETS measurement as a change in centimeters (cm). This is a longitudinal assessment of balance following surgical intervention for CSM.
Time Frame: Pre-surgery compared to 2 weeks, 6 weeks, and 6 months post-surgery VETS factors. The Post-surgery endpoints are normally scheduled clinical follow ups.
Population: Subjects were gradually lost to follow-up, leading to a decline in the number of participants analyzed in later sessions.
Measure: Mean (Standard Deviation); unit: CM
Groups:
- Cervical Spondylotic Myelopathy (CSM) Group: Veterans with CMS. CMS is a degenerative cervical myelopathy, encapsulates a cascade of events leading to significant degenerative changes in discs, formation of osteophytes, facet hypertrophy, calcification of the posterior longitudinal ligament and ligamentous flavum with resultant canal stenosis and segmental instability.
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group
Number analyzed (Participants) | 6
CM
  EO Firm PreOp | 11 (27.1)
  EC Firm PreOp | 13 (15.4)
  DYN Firm PreOp | 48.4 (51.1)
  EO Foam PreOp | 19.1 (20.3)
  EC Foam PreOp | 44 (32.7)
  DYN Foam PreOp | 70.7 (47.7)
  EO Firm 2Weeks: number analyzed (Participants) | 5
  EO Firm 2Weeks | 5.6 (4.3)
  EC Firm 2Weeks: number analyzed (Participants) | 5
  EC Firm 2Weeks | 9.4 (8.5)
  DYN Firm 2Weeks: number analyzed (Participants) | 5
  DYN Firm 2Weeks | 11.2 (7)
  EO Foam 2Weeks: number analyzed (Participants) | 5
  EO Foam 2Weeks | 9.8 (7)
  EC Foam 2Weeks: number analyzed (Participants) | 5
  EC Foam 2Weeks | 44.3 (28.7)
  DYN Foam 2Weeks: number analyzed (Participants) | 5
  DYN Foam 2Weeks | 63.5 (39.6)
  EO Firm 6Weeks: number analyzed (Participants) | 4
  EO Firm 6Weeks | 7.2 (9.8)
  EC Firm 6Weeks: number analyzed (Participants) | 4
  EC Firm 6Weeks | 15.6 (22.1)
  DYN Firm 6Weeks: number analyzed (Participants) | 4
  DYN Firm 6Weeks | 15.4 (15.1)
  EO Foam 6Weeks: number analyzed (Participants) | 4
  EO Foam 6Weeks | 12.2 (7.5)
  EC Foam 6Weeks: number analyzed (Participants) | 4
  EC Foam 6Weeks | 37.6 (31)
  DYN Foam 6Weeks: number analyzed (Participants) | 4
  DYN Foam 6Weeks | 88.5 (68.7)
  EO Firm 6Months: number analyzed (Participants) | 3
  EO Firm 6Months | 5 (5.4)
  EC Firm 6Months: number analyzed (Participants) | 3
  EC Firm 6Months | 12 (15.1)
  DYN Firm 6Months: number analyzed (Participants) | 3
  DYN Firm 6Months | 24.7 (33.8)
  EO Foam 6Months: number analyzed (Participants) | 3
  EO Foam 6Months | 13.5 (6.1)
  EC Foam 6Months: number analyzed (Participants) | 3
  EC Foam 6Months | 41.4 (19.1)
  DYN Foam 6Months: number analyzed (Participants) | 3
  DYN Foam 6Months | 62.9 (38.1)

3. Secondary Outcome: Nurick Scale
Description: The Nurick scale is a 6-grade ordinal scale assessing gait impairment, with grades ranging from 0 (signs and symptoms of root involvement but no evidence of spinal cord disease) to 5 (chair bound or bedridden). The aggregate value of the Nurick scale will be related to posturography. Classification Scheme:
  * Grade 0: signs or symptoms of root involvement but without evidence of spinal cord disease
  * Grade 1: signs of spinal cord disease but no difficulty in walking.
  * Grade 2: slight difficulty in walking which does not prevent full-time employment
  * Grade 3: difficulty in walking which prevented full time employment or the ability to do all housework, but which was not so severe as to require someone else's help to walk
  * Grade 4: able to walk only with someone else's help or with the aid of a frame.
  * Grade 5 : chairbound or bedridden.
Time Frame: PreSurgery compared to otherwise healthy Veterans
Population: The investigators did not recruit any controls as we could not run participants who did not already have a clinical appointment, due to COVID restrictions
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group | Healthy Controls
Number analyzed (Participants) | 6 | 0
Units on a scale | 2 (.89) |

4. Secondary Outcome: Neck Disability Index (NDI)
Description: NDI is related to VETS posturography to determine sensitivity of standing posture to degree of disability. The NDI is a 10-item questionnaire addressing function activities (personal care, lifting, reading, work, driving, sleeping, and recreation), pain intensity, concentration, and headache. For each item, patients make their ratings on a 6-point Likert scale with values 0 = no disability and 5 = complete disability. Summed scores for each category are multiplied by 2 to give a total NDI score ranging from 0-100. Score: /50 Transform to percentage score x 100 = %points. Scoring: Example:16 (total scored)50 (total possible score) x 100 = 32% If one section is missed or not applicable the score is calculated: 16 (total scored)45 (total possible score) x 100 = 35.5% Minimum Detectable Change (90% confidence): 5 points or 10 %points
Time Frame: PreSurgery compared to otherwise healthy Veterans
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group | Healthy Controls
Number analyzed (Participants) | 6 | 0
Units on a scale | 59.5 (17.5) |

5. Secondary Outcome: Short Form-36 Version 2 (SF-36v2)
Description: The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). The SF-36 offers a choice of recall format at a standard (4 week) or acute (1 week) time frame. Likert scales and yes/no options are used to assess function and well-being on this 36-item questionnaire. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Time Frame: PreSurgery compared to otherwise healthy Veterans
Population: Healthy controls could not be recruited because of COVID restrictions
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group | Healthy Controls
Number analyzed (Participants) | 6 | 0
Units on a scale | 44.1 (21.1) |

6. Secondary Outcome: EC FIRM/EO FIRM Ratio
Description: From the VETS, a ratio corresponding to the Rhomberg ratio of COP sway will be used to determine the degree static posture depends on visual input. The Romberg test used in posturography compares postural sway in eyes open (EO) and eyes closed (EC) conditions. The Romberg ratio was calculated in the traditional manner, i.e. EC/EO. The ensuing Romberg ratio (EC/EO) is used to assess visual dependency in postural stability. Higher Romberg ratios reflect greater instability with closed eyes, ( a greater amount of postural sway during eyes closed) whereas a ratio < 1 indicates higher stability in the EC versus EO condition.
Time Frame: PreSurgery
Measure: Mean (Standard Deviation); unit: COP sway ratio
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group
Number analyzed (Participants) | 6
COP sway ratio | 1.56 (1.03)

7. Secondary Outcome: EO FOAM/EO FIRM
Description: From the VETS, a ratio of COP sway will be used to determine the degree static posture is affected by reduced proprioception.
Time Frame: PreSurgery compared to otherwise healthy Veterans
Population: The investigators could not recruit controls due to COVID restrictions
Measure: Mean (Standard Deviation); unit: COP sway ratio
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group | Healthy Controls
Number analyzed (Participants) | 6 | 0
COP sway ratio | 2.92 (3.17) |

8. Secondary Outcome: EC FOAM/EO FOAM Ratio
Description: From the VETS, a ratio of COP sway will be used to determine the degree of loss of visual information. Loss of visual information compounds reduced proprioceptive ability in static balance.
Time Frame: PreSurgery compared to otherwise healthy Veterans
Population: Could not recruit controls due to COVID restrictions
Measure: Mean (Standard Deviation); unit: COP sway ratio
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group | Healthy Controls
Number analyzed (Participants) | 6 | 0
COP sway ratio | 8.43 (11.8) |

9. Secondary Outcome: DYN FOAM/DYN FIRM Ratio
Description: From the VETS, a ratio of COP sway will be used to determine how roll vection is induced by loss of proprioception.
Time Frame: PostSurgery compared to otherwise healthy Veterans compared to otherwise healthy Veterans
Population: Could not recruit controls due to COVID restrictions. Only 4 CSM participants were analyzed compared to the 6 anticipated due to data capture failure in 2 participants during DYN Foam condition and facility entrance policies restricted patient flow for the remainder of the study. Three of them had incomplete trial sessions, but this does not affect overall calculation as this was taken into consideration.
Measure: Mean (Standard Deviation); unit: COP Sway ratio
Arm/Group | Cervical Spondylotic Myelopathy (CSM) Group | Healthy Controls
Number analyzed (Participants) | 4 | 0
COP Sway ratio | 8.7 (13.76) |

10. Secondary Outcome: DYN FIRM/ EO FIRM Ratio
Description: From the VETS, a ration of COP sway to determine the degree roll vection is induced.
Time Frame: PreSurgery compared to otherwise healthy Veterans
Population: Could not recruit controls due to COVID restrictions
Measure: Mean (Standard Deviation); unit: COP Sway ratio
Arm/Group | Cervical Spondylotic Myelopathy (CSM) | Healthy Controls
Number analyzed (Participants) | 6 | 0
COP Sway ratio | 6.49 (6.62) |

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time of study entry until the end of study participation, and average of 6 months
Arm/Group | Cervical Spondylotic Myelopathy (CSM)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
COVID significantly disrupted our ability to complete the study. Scheduling for CSM surgery was drastically impacted by COVID and never returned to Pre-COVID format. Some subjects recruited before COVID could not be followed up due to a ban on research. We were also unable to recruit controls because our VA only permitted research appointments for individuals who were already coming to the VA for a medical appointment (e.g. surgical follow-up).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT03810781/Prot_SAP_000.pdf